CLINICAL TRIAL: NCT03653936
Title: Neuro-ocular Baselines in a Sports Setting: Feasibility Study for Head and Intraocular Trauma Test (HITT) Device for Potential Detection of Brain Dysfunction
Brief Title: Neuro-ocular Baselines in a Sports Setting
Acronym: KY
Status: Completed | Type: Observational
Sponsor: Rebiscan, Inc. (Industry)
Collaborators: BlueGrass Orthopaedics Surgery & Hand Care (Unknown)
Responsible Party: Sponsor
Other Study IDs: Rebiscan-005
Record Dates: First submitted 2018-08-28; First posted 2018-08-31 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Wave Form Signals Coming From the Eye in a Healthy Cohort

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: HITT device — Rebion has developed a noninvasive, handheld device that uses retinal polarization scanning (RPS) to rapidly assess eye fixation and retinal integrity in adults and children. RPS can automatically detect the fixation of the human eye with proprietary technology that uses a scanned annulus of polarized laser light to create a signature that confirms central fixation within seconds. RPS requires no calibration or imaging, and eye movement recordings are not required. The HITT device is a repurposed Pediatric Vision Scanner (PVS), Rebion's first commercial product which has passed all applicable safety and performance standards.

SUMMARY:
Rebion (Rebiscan, Inc) has developed a noninvasive, handheld device that uses retinal birefringence scanning (RBS) to rapidly assess eye fixation and retinal integrity in adults and children. The proprietary technology uses a scanned annulus of polarized laser light to create a signature that confirms central fixation within seconds. The project described herein aims to provide accurate assessment of brain dysfunction in TBI (Traumatic Brain Injury) patients through the use of the developed device, which is called the Head and Intraocular Trauma Test (HITT) device.

ELIGIBILITY:
Inclusion Criteria:

* Student-athletes who present to schools affiliated with the Bluegrass Sports Clinica
* Engaged in sports
* Older or equal to 11 years of age, and less than 21 years of age.
* Provide informed consent; youths must have their parents sign the informed consent document. Children will be presented with a written assent statement and that they will be asked to sign the assent document.

Exclusion Criteria:

* Catastrophic polytrauma that would interfere with follow-up and outcome assessment
* Amblyopia/strabismus
* Pregnancy in female subjects
* Any injury to eye including, puncture, scratch, occlusion, fracture to orbital socket (or any fracture to face that would negatively impact eye movement/vision) that would interfere with ability to complete study-device assessment.
* History of poor vision prior to injury (Visual acuity worse than 20/40 in either eye)
* Intoxication or chemical impairment at time of examination (upon initial presentation)

Ages: 11 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Cohort study of individuals tested with the Rebion device followed by SCAT3 examination. Two data sets will be taken and compared: a cohort with non-contact sport athletes (swimmers, tennis, track) and a cohort of contact sport athletes (lacrosse, spring football, and spring soccer).
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Capturing of wave forms from the eye | Screenings will be performed during a normally scheduled visit to the sports facility by the research group enrolling in the study
  Screening device will provide a wave form calculation of light reflecting off patient's eye

CONTACTS AND LOCATIONS:
Overall Officials: Harry Lockstadt, MD, Principal Investigator — Bluegrass Orthopaedics
Locations (1):
- BlueGrass Orthopaedics, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Undecided